CLINICAL TRIAL: NCT02546310
Title: Interventional, Randomised, Double-blind, Parallel-group, Placebo-controlled, Phase 1, Exploratory Study Investigating the Effects of HTL0009936 on Cognition and BOLD fMRI Signals in Healthy Elderly Subjects
Brief Title: Phase 1 Study Investigating Effects of HTL0009936 on Cognition and BOLD fMRI Signals in Healthy Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nxera Pharma UK Limited (Industry)
Collaborators: P1vital Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 9936-103
Record Dates: First submitted 2015-09-01; First posted 2015-09-10 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- HTL0009936 high dose (Experimental): high dose infusion
  Interventions: Drug: HTL0009936
- HTL0009936 low dose (Experimental): low dose infusion
  Interventions: Drug: HTL0009936
- HTL0009936 matching placebo (Placebo Comparator): matching infusion
  Interventions: Drug: HTL0009936 matching placebo

INTERVENTIONS:
Drug: HTL0009936
  Arms: HTL0009936 high dose; HTL0009936 low dose
Drug: HTL0009936 matching placebo
  Arms: HTL0009936 matching placebo

SUMMARY:
To determine if treatment with HTL0009936 will lead to changes in neural activity, measured using the fMRI BOLD signal and ASL, in brain areas that are associated with spatial and working memory, learning and executive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history, physical examination, vital signs, 12-lead ECG, haematology, blood chemistry, urinalysis and a pre-study psychological assessment.
* Mini Mental State Examination (MMSE) Score of ≥24.
* Intermediate or extensive metaboliser as determined by CYP2D6 genotype.
* Fluent English speaker.
* Right-handed.
* Not a regular smoker

Exclusion Criteria:

* Recreational drug use within 3 months prior to Screening Visit.
* Positive alcohol breath test.
* Positive urine drug screen.
* Consumption of large amounts of caffeinated drinks.
* Consumption of any food or any drinks containing cranberry, pomegranate, star fruit, grapefruit, pomelos, exotic citrus fruits or Seville oranges.
* Ultra-rapid or poor metabolizer as determined by CYP2D6 genotype.
* By self-report, taking two or more daytime naps per week which in the opinion of the investigator is likely to interfere with the ability of the subject to complete the study procedures.
* History of, or presents (in the opinion of the Investigator) with, significant neurological or psychiatric conditions.
* Personal or family history of congenital long QT syndrome or sudden death.
* Concomitant use of drugs that are metabolised by and/or are inhibitors of CYP2D6.
* Concomitant use of drugs that are substrates for the organic cation transporter 2.
* History of significant claustrophobia.
* Fulfils any of the MRI contraindications on the standard site radiography screening questionnaire (e.g. history of surgery involving metal implants).

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Blood oxygen level dependent (BOLD) signal in functional Magnetic Resonance Imaging (fMRI) of the brain areas associated with cognitive tasks | Day 1

SECONDARY OUTCOMES:
BOLD signal in fMRI in other brain regions involved in the regulation of cognitive processes during cognitive tasks | Day 1
cerebral blood flow, assessed using Arterial Spin Labelling (ASL) | Day 1
adverse events | Day 1
blood pressure | Day 1
12-lead electrocardiogram | Day 1

OTHER OUTCOMES:
event related potentials | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Neuroscience and Psychiatry Unit, Manchester, United Kingdom